CLINICAL TRIAL: NCT06033482
Title: A Single Center, Prospective Study on the Possible Range of No.12a Lymph Node Dissection of Locally Advanced Gastric Cancer
Brief Title: The Possible Range of No.12a Lymph Node Dissection of Locally Advanced Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: E20230548
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Gastric Cancer; No.12a Lymph Node Dissection
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: The reasonable range of No.12a lymph node dissection — The lymph node overlying the proper hepatic artery is defined as No.12aa. The lymph node overlying the left side of the portal vein is defined as No.12av. Observation of lymph node metastasis rates in two groups.

SUMMARY:
The main purpose of this study is to evaluate the reasonable range of No.12a lymph node dissection of locally advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤ 75 years of age; Preoperative gastric cancer patients with pathologically confirmed; Had been treated with Radical resection (D2, R0) of gastric cancer (Lymph node≥16); Willing and able to comply with the program during the study period; Physical condition and organ function allows to tolerable abdominal surgery; Written informed consent provided; Under radical laparoscopic distal subtotal gastrectomy With more than a 6-month life expectancy; No other serious concomitant diseases; Sufficient organ functions; No previous history of chemotherapy or radiotherapy; Clinical stage: T2-4aNxM0; Karnofsky performance status (KPS)>60; Eastern Cooperative Oncology Group Performance Status (ECOG): 0-1.

Exclusion Criteria:

* Pregnancy or breast feeding; Patients with Serious liver disease (such as cirrhosis, etc.), kidney disease, respiratory disease or uncontrolled diabetes, hypertension and other chronic systemic diseases, heart disease with Clinical symptoms, such as congestive heart failure, coronary heart disease symptoms, drug is difficult to control arrhythmia, hypertension, or six months had a myocardial infarction attack, or cardiac insufficiency; Organ transplantation patients need immunosuppressive therapy; Severe recurrent infections were not controlled or with other serious concomitant diseases; Patients got other primary malignant tumors (except curable skin basal cell carcinoma and cervical cancer in situ) except gastric cancer within 5 years; Psychiatric disease which require treatment; Have the history of organ transplantation; Within 6 months before study starts and in the process of this study, patients participate in other clinical researches.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients with advanced gastric cancer，underwent radical laparoscopic distal gastrectomy. Observation of lymph node metastasis in different No.12a subgroups.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The lymph node metastasis rates in No.12aa and No.12av groups. | 100 cases enrolled within 1 year
  Observation of lymph node metastasis in different No.12a subgroups12 years

CONTACTS AND LOCATIONS:
Overall Officials: Bin Ke, MD, Study Director — Department of Gastric cancer, Tianjin Medical University Cancer Institute & Hospital; Peng Ru Zhang, MD, Study Director — Department of Gastric cancer, Tianjin Medical University Cancer Institute & Hospital
Locations (1):
- Department of Gastric cancer, Tianjin Medical University Cancer Institute & Hospital,, Tianjin, None Selected, China

IPD SHARING:
Plan to Share IPD: No